CLINICAL TRIAL: NCT02053168
Title: A Prospective, Multicenter All Comers Study of a Novel Resorbable Mesh (Phasix Mesh) for Ventral or Incisional Hernia Repair
Brief Title: A Prospective, Multicenter All Comers Study of Phasix Mesh for Ventral or Incisional Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVL-HE-015
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Ventral Hernia; Incisional Hernia
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resorbable Mesh (Other): Phasix Mesh
  Interventions: Device: Resorbable Mesh

INTERVENTIONS:
Device: Resorbable Mesh — Phasix Mesh

SUMMARY:
Collect data on safety, performance, and effectiveness of Phasix Mesh in subject requiring primary ventral and incisional hernias.

DETAILED DESCRIPTION:
Pilot Study of patients across all wound classes for recurrence

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's legally authorized representative must be willing to give written informed consent
* Subject must be diagnosed with ventral or incisional hernia
* Subject must be willing to undergo open ventral hernia repair and be able to undergo all other study procedures as outlined in this protocol.

Exclusion Criteria:

* Subject is an active smoker (if attempts to quit smoking within two weeks of surgery have failed and the patient is still an active smoker at the time of surgery).
* Subject's hernia has recurred four or more times.
* Subject's body mass index (BMI) >40 kg/m2.
* Subject has peritonitis.
* Subject is on or suspected to be placed on chemotherapy medications during any part of the study.
* Chronic steroid use or immunosuppression drugs (> 6 months).
* Subject has cirrhosis, and/or ascites.
* Subject is American Society of Anesthesiology Class 4 or 5.
* Subject is pregnant or planning to become pregnant during the course of the study.
* Subject is known to be infected with human immunodeficiency virus (HIV).
* Subject has a life expectancy of less than 2 years at the time of enrollment.
* Subject has been treated with an investigational product in the past 30 days.
* Subject is part of the site personnel directly involved with this study
* Subject has a known allergy to tetracycline hydrochloride or kanamycin sulfate, the test device or its component materials.
* Subject has any condition that in the opinion of the Investigator would preclude the use of the study device, or preclude the subject from completing the follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02; Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Novitsky, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (6):
- United States (6):
  - Beverly Hills Hernia Center, Beverly Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Florida Hospital Celebration Health, Celebration, Florida
  - Methodist Physicians Clinic, Omaha, Nebraska
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon Health and Sciences University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 33 subjects enrolled, 8 were not treated with the study device: a contraindication to the placement of mesh was present in 4 subjects; complete removal of existing mesh from a prior hernia repair (in the same affected area) was not possible in 3 subjects; and 1 subject had an active or latent systemic infection.
Period: Overall Study
Arm/Group | Resorbable Mesh
Started | 25
Completed | 22
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (17.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Weight [Mean (Standard Deviation); unit: kg] | 84.3 (17.16)
Height [Mean (Standard Deviation); unit: cm] | 166.9 (7.53)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (5.81)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hernia Recurrence
Description: A recurrent hernia was defined as any hernia identified or confirmed by the investigator, during any study follow-up visit, in approximately the same position as the hernia repaired in the study procedure. Potential hernias identified via incidental magnetic resonance imaging (MRI) or computed tomography (CT) scan were evaluated by the operating surgeon for clinical significance and confirmation of hernia recurrence.
Time Frame: 1 Month, 3 Months, 6 Months, 12 Months, 18 Months, 24 Months, >24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
Participants
  1 Month | 0
  3 Months | 0
  6 Months | 0
  12 Months | 1
  18 Months | 0
  24 Months | 0
  >24 Months | 1
  Post Op to End of Study | 2

2. Secondary Outcome: Number of Participants With Device Related Adverse Events
Description: In this study, a device-related adverse event is defined as any undesirable clinical event occurring in the abdominal space including the lower abdominal, inguinal and pubic regions (including the skin), as well as any other undesirable clinical events judged to be related to the study device or surgical procedure regardless of anatomical region.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
Participants | 1

3. Secondary Outcome: Carolinas Comfort Scale (CCS) Total Score - Change From Baseline
Description: The Carolinas Comfort Scale is a short, hernia-specific 8-category questionnaire designed to measure patient perception of symptoms and patient satisfaction with a scale from 0 (no symptoms) to 5 (disabling symptoms). The change was calculated as the mean value at 24 months minus the mean value at baseline.
Time Frame: Baseline and 24 months postoperative
Population: All participants with non-missing values at both baseline and respective post procedure assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 8
units on a scale | -1.1 (1.12)

4. Secondary Outcome: Short Form (SF)-12 Version 2 - Physical Component Summary (Change From Baseline)
Description: Short Form (SF)-12 Version 2 is a multipurpose, 12-item health survey that measures seven domains of health: general health, physical functioning, role limitations due to physical health (role-physical), role limitations due to emotional problems (role-emotional), bodily pain, vitality and mental health, and social functioning. It yields two summary measures of physical and mental health: the physical component summary (PCS) and mental component summary (MCS). The scores range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The change was calculated as the mean value at 24 months minus the mean value at baseline.
Time Frame: Baseline and 24 months postoperative
Population: All participants with non-missing values at both baseline and respective post procedure assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 21
units on a scale | -5.3 (9.98)

5. Secondary Outcome: Short Form (SF)-12 Version 2 - Mental Component Summary (Change From Baseline)
Description: Short Form (SF)-12 Version 2 is a multipurpose, 12-item health survey that measures seven domains of health: general health, physical functioning, role limitations due to physical health (role-physical), role limitations due to emotional problems (role-emotional), bodily pain, vitality and mental health, and social functioning. It yields scale scores for each of these seven health domains, and two summary measures of physical and mental health: the physical component summary (PCS) and mental component summary (MCS). The scores range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The change was calculated as the mean value at 24 months minus the mean value at baseline.
Time Frame: Baseline and 24 months postoperative
Population: All participants with non-missing values at both baseline and respective post procedure assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 21
units on a scale | -9.4 (9.21)

6. Secondary Outcome: Surgical Procedure Time
Description: Measured from incision to closure (skin to skin).
Time Frame: Duration of index procedure (mean of 242.5 mins)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
minutes | 242.5 (132.2)

7. Secondary Outcome: Length of Hospital Stay
Description: Measured from end of index procedure to hospital discharge
Time Frame: 10 Months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
days | 5.0 (4.04)

8. Secondary Outcome: Number of Study Related Post Operative Surgical Procedures
Time Frame: 24 Months
Measure: Number; unit: events
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
events | 7

9. Secondary Outcome: Number of Study Related Post Operative New Hospital Admissions
Time Frame: 24 Months
Measure: Number; unit: events
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
events | 5

10. Secondary Outcome: Number of Related Post-operative Visits Unrelated to Standard of Care
Time Frame: 24 Months
Measure: Number; unit: events
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
events | 8

11. Secondary Outcome: Incidence of Seroma
Time Frame: 24 Months
Measure: Number; unit: events
Arm/Group | Resorbable Mesh
Number analyzed (Participants) | 25
events | 1

ADVERSE EVENTS:
Time Frame: Up to 24 months post index procedure
Arm/Group | Resorbable Mesh
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 6/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resorbable Mesh (N=25)
Superficial surgical site infection (Infections and infestations) | 1 (2)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (2)
Seroma (General disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1)
Myocardial hypoxia (Cardiac disorders) | 1 (1)
Abdominal wall wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resorbable Mesh (N=25)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-08-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT02053168/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT02053168/SAP_001.pdf